CLINICAL TRIAL: NCT04949958
Title: Effects of Exercise Based Manual on Biochemical, Cardiorespiratory and Physical Parameters in Sedentary Prediabetic Population
Brief Title: Effects of Exercise Based Manual in Sedentary Prediabetic Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: REC/Lhr/21/1103 Sana Hafeez
Record Dates: First submitted 2021-06-26; First posted 2021-07-02 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: PreDiabetes
Keywords: Prediabetic; Exercise intervention; Biochemical parameters; Cardiorespiratory parameters; Physical parameters
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Intervention Model Description: Experimental: Exercise Based Manual (Supervised) Supervised exercise based Manual (exercise & Educational Component) for 3 days / week for 16 weeks. Each session will comprise of 60 minutes of combination of different exercises including warm up and rest interval
  Experimental: Exercise Based Manual (Home Based) Home Based- Exercise Manual (Exercise & Educational Component) for 16 weeks. Subject will be asked to maintain a regular exercise and dietary education to ensure adherence to the program
  Placebo Comparator: Control Age matched Control Group followed for 16 weeks with General Advise to be active.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: Exercise Based Manual (Supervised) (Experimental): Supervised Exercises with exercise based Manual (exercise & Educational Component) for 3 days / week for 16 weeks. Each session will comprise of 60 minutes of different type of exercises including warm up and rest interval
  Interventions: Other: Exercise Based Manual (Supervised)
- Experimental: Exercise Based Manual (Home Based) (Experimental): Experimental: Exercise Based Manual (Home Based) Home Based- Exercise Manual (Exercise & Educational Component) for 16 weeks. Subject will be asked to maintain a regular exercise.
  Interventions: Other: Exercise Based Manual (Home Based)
- Placebo Comparator: Control (Placebo Comparator): Age matched Control Group followed for 16 weeks with General Advise to active
  Interventions: Other: Control

INTERVENTIONS:
Other: Exercise Based Manual (Supervised) — Exercise Based Manual for Pre Diabetic subjects will consist of two components; Exercise, Exercise and Education. The exercise will be supervised while other component will be home based.
  Arms: Experimental: Exercise Based Manual (Supervised)
Other: Exercise Based Manual (Home Based) — Exercise Based Manual for Pre Diabetic subjects will consist of two components; Exercise and Education. All two components will be home based.
  Arms: Experimental: Exercise Based Manual (Home Based)
Other: Control — General advice to be active
  Arms: Placebo Comparator: Control

SUMMARY:
The prediabetes is a state in which fasting blood glucose level ranges between 100-126mg/dl or HbA1C ranges between 5.7-6.4mmol. People with prediabetes have 74 percent chance of progression to develop Type 2 diabetes mellitus. However, by lifestyle intervention, Type 2 Diabetes mellitus may be effectively avoided or delayed. The improvement in lifestyle is involving the physical activity of at least 150mins per week lowered the rate of T2DM in people with prediabetes by 58 percent. There are several risk factors for the development of type 2 diabetes mellitus, but obesity and lack of physical activity are major risk factors that cause type 2 diabetes mellitus in prediabetic populations. Diet and exercise are the first line treatment for sedentary prediabetics. Both independent and combined effect of diet and exercise can reduce the incidence of T2DM, glycemic control and weight loss in adults with prediabetics

DETAILED DESCRIPTION:
The most alarming public health issues of the 21st century is epidemic of diabetes especially in lower middle-income countries. There will be a 67 percent raise in prevalence of diabetes from 2010 to 2030 .With up to half of deaths occurring in people under the age of 60 is due to diabetes as T2DM is among the top ten causes of death.According to American Diabetic Association, if Fasting blood glucose level falls between <100mg/dl or HbA1C falls between <5.7% then person has normal blood sugar level if Fasting blood glucose level falls between 100-125mg/dl or HbA1C falls between 5.7%-6.4% then person is diagnosed as prediabetic and if value of fasting blood glucose level falls between 126-200mg/dl and HbA1C more than 6.5% then person is diagnose as Type 2 Diabetes mellitus.

Prediabetes is a state in which the body can maintain blood glucose level but impaired insulin sensitivity is still present.Worldwide there is a 74 percent chance of progression of prediabetes into Type 2 Diabetes Mellitus. Strategies for prevention of T2DM are highly recommended for sedentary population.There are now estimated 38 million adults living with diabetes around the world. The main cause of premature death in the world with ration of every 6 into 10 due to the effects of diabetes and diabetes-related complications.

Pakistan is now in the top 10 countries with increase in the incidence of diabetes. According to WHO, around 19 million people are diagnosed with diabetes and 10 million people are diagnosed as prediabetics. An estimated 463 million adults worldwide live with diabetes and 55 million live with prediabetes. However there are some risk factors for T2DM that can be modifiable including obesity, metabolic syndrome characteristics (abdominal obesity, elevated triglycerides, low density lipoprotein), high blood pressure and elevated plasma glucose, insulin resistance, sedentary lifestyle Exercise intervention requires repetitive body movements performed to enhance or sustain one or more physical fitness components such as aerobic ability, muscle strength and endurance, flexibility. Sedentary lifestyle is associated with an increased risk of death, cardiovascular disease and increase the incidence of T2DM which is mostly recognized in young adult population.Physical exercise facilitates improved functioning of the human body. Regular exercise enhances insulin sensitivity thus helping to avoid diabetes.Exercise training is known to increase the absorption of insulin-mediated skeletal muscle glucose and blood flow to limbs thus leading to reduction in glycemic control in diabetic population.

ELIGIBILITY:
Inclusion Criteria:

* Serum glucose test indicating prediabetic (HbA1c level of 5.7% - 6.4% or fasting plasma glucose of 100 - 12
* Sedentary Subjects (<150 min/week or <600 MET-min/week on IPAQ Urdu Version)

Exclusion Criteria:•

* History of type 2 diabetes mellitus or newly diagnosed diabetes within last 6 months
* BMI under 18.5 and more 30
* Persons involve in other weight management program,
* History of taking any herbal medications to control the weight
* Clinical history of cardiovascular diseases occurred within the past six months
* Pregnancy

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c Test (HbA1C0 | 16 week
  Hemoglobin A1c Test tells you average level of blood sugar over the past 2 to 3 months.The normal range for the hemoglobin A1c level is between 4% and 5.6% and readings will be taken at baseline,8th week and 16 week.
Fasting blood Glucose(FBG) | 16 weeks
  This test checks your fasting blood sugar levels. Fasting means after not having anything to eat or drink (except water) for at least 8 hours before the test. Normal value will be less than 100 mg/dl and Prediabetes value 100 mg/dl to 125 mg/dl.Reading will be taken after 8 hour fasting. Readings will be taken at baseline,8th week and 16 week
Homeostasis model assessment of β-cell function(HOMA-β) | 16 weeks
  The homeostasis model assessment of β-cell function (HOMA-β) is an index of insulin secretory function derived from fasting plasma glucose and insulin concentrations.It is calculated by using the following formula: 360 x fasting insulin (μU/mL) / (fasting glucose (mg/dL) - 63).Sample will be taken from intravenous blood sample & readings will be taken at baseline and at 16 weeks.
Homeostatic Model Assessment for Insulin Resistance(HOMA-IR) | 16 weeks
  Homeostatic model assessment (HOMA) is a method for assessing β-cell function and insulin resistance (IR) from basal (fasting) glucose and insulin or C-peptide concentrations. Healthy Range: 1.0 (0.5-1.4).Less than 1.0 means you are insulin-sensitive which is optimal. Above 1.9 indicates early insulin resistance. sample will be taken from intravenous blood sample & readings will be taken at baseline and at 16 weeks.
low-density lipoproteins(LDL) | 16 weeks
  low-density lipoproteins sometimes called the "bad" cholesterol Value Less than 100mg/dL is Optimal, value 100-129mg/dL Near optimal/above optimal,Value 130-159 mg/dL Borderline high. Reading will be taken at baseline,8th week and at 16 weeks of intervention.
high-density lipoproteins( HDL) | 16 weeks
  high-density lipoproteins sometimes called the "good" cholesterol.HDL that falls within the range of 40 to 59 mg/dL is normal. Readings will be taken at baseline,8th week and 16 weeks of intervention.
Triglycerides | 16 weeks
  Triglycerides are a type of fat (lipid) found in your blood. Normal triglyceride levels in the blood are less than 150 mg per deciliter (mg/dL). Readings will be taken at baseline,8th week and 16 weeks of intervention.
Maximal oxygen consumption( VO2max) | 16 weeks
  the maximum or optimum rate at which the heart, lungs, and muscles can effectively use oxygen during exercise, used as a way of measuring a person's individual aerobic capacity.A good VO2 max for a male is 42.5-46.4 mL/kg/min, while a good value for a female is 33.0-36.9 mL/kg/min.Readings will be taken at baseline,8th week and 16 weeks of intervention.
Rate of perceived exertion( PRE) | 16 weeks
  The RPE scale is used to measure the intensity of your exercise. The RPE scale runs from 0 - 10. Readings will be taken at baseline,8th week and 16 weeks of intervention.
Baseline Dyspnea Index(BDI) | 16 weeks
  Baseline Dyspnea Index (BDI) measures the severity of dyspnea at the baseline Readings will be taken at baseline,8th week and 16 weeks of intervention.
weight in kilograms | 16 weeks
  Weight (symbolized w ) is a quantity representing the force exerted on a particle or object by an acceleration field, particularly the gravitational field of the Earth at the surface.Readings will be taken at baseline,8th week and 16 weeks of intervention.
Body mass index (BMI) | 16 weeks
  is a measure of body fat based on height and weight that applies to adult men and women. Below 18.5 is Underweight,18.5-24.9 is Normal,25.0-29.9 is Overweight, 30.0 and Above is Obese. Readings will be taken at baseline,8th week and 16 weeks of intervention.
waist circumference | 16 weeks
  Waist circumference is the measurement taken around the abdomen at the level of the umbilicus (belly button). For best health, waist should be less than 40 inches around for men, and less than 35 inches for women. Readings will be taken at baseline,8th week and 16 weeks of intervention with use of inelastic measuring tape.
waist to hip ratio (WHR) | 16 weeks
  Waist too hip ratio is a quick measure of fat distribution that may help indicate a person's overall health. A healthy WHR is: 0.9 or less in men. 0.85 or less for women. Readings will be taken at baseline,8th week and 16 weeks of intervention with use of inelastic measuring tape.
Body fat percentage | 16 weeks
  body fat percentage as just one way to assess and monitor your weight and overall body composition.Men Women Average value for men is18%-24% and foe women is 25%-31%.Value for Obese men is 25% and higher, for obese women is 32% and higher. Readings will be taken at baseline,8th week and 16 weeks of intervention with use of body fat analyzer.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil ur Rehman, PhD, Study Chair — Riphah International University
Locations (1):
- Riphah Rehabiliation Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rowan CP, Riddell MC, Gledhill N, Jamnik VK. Aerobic Exercise Training Modalities and Prediabetes Risk Reduction. Med Sci Sports Exerc. 2017 Mar;49(3):403-412. doi: 10.1249/MSS.0000000000001135. PMID 27776003
- [Background] Williams AN, Konopken YP, Keller CS, Castro FG, Arcoleo KJ, Barraza E, Patrick DL, Olson ML, Shaibi GQ. Corrigendum to 'Culturally-grounded diabetes prevention program for obese Latino youth: Rationale, design, and methods☆'' [Contemp. Clin. Trials 54 (2017) 68-76]. Contemp Clin Trials. 2018 Aug;71:205. doi: 10.1016/j.cct.2018.06.014. Epub 2018 Jul 7. No abstract available. PMID 30064689
- [Background] Aguiar EJ, Morgan PJ, Collins CE, Plotnikoff RC, Callister R. Efficacy of interventions that include diet, aerobic and resistance training components for type 2 diabetes prevention: a systematic review with meta-analysis. Int J Behav Nutr Phys Act. 2014 Jan 15;11:2. doi: 10.1186/1479-5868-11-2. PMID 24423095
- [Background] Barengo NC, Tuomilehto J. Diabetes: exercise benefits in type 2 diabetes mellitus. Nat Rev Endocrinol. 2012 Nov;8(11):635-6. doi: 10.1038/nrendo.2012.182. Epub 2012 Oct 2. No abstract available. PMID 23032182
- [Background] Rhodes EC, Chandrasekar EK, Patel SA, Narayan KMV, Joshua TV, Williams LB, Marion L, Ali MK. Cost-effectiveness of a faith-based lifestyle intervention for diabetes prevention among African Americans: A within-trial analysis. Diabetes Res Clin Pract. 2018 Dec;146:85-92. doi: 10.1016/j.diabres.2018.09.016. Epub 2018 Sep 28. PMID 30273708
- [Background] Jensen MD, Ryan DH, Apovian CM, Ard JD, Comuzzie AG, Donato KA, Hu FB, Hubbard VS, Jakicic JM, Kushner RF, Loria CM, Millen BE, Nonas CA, Pi-Sunyer FX, Stevens J, Stevens VJ, Wadden TA, Wolfe BM, Yanovski SZ; American College of Cardiology/American Heart Association Task Force on Practice Guidelines; Obesity Society. 2013 AHA/ACC/TOS guideline for the management of overweight and obesity in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and The Obesity Society. J Am Coll Cardiol. 2014 Jul 1;63(25 Pt B):2985-3023. doi: 10.1016/j.jacc.2013.11.004. Epub 2013 Nov 12. No abstract available. PMID 24239920
- [Background] Kosaka K, Noda M, Kuzuya T. Prevention of type 2 diabetes by lifestyle intervention: a Japanese trial in IGT males. Diabetes Res Clin Pract. 2005 Feb;67(2):152-62. doi: 10.1016/j.diabres.2004.06.010. PMID 15649575
- [Background] Pan XR, Li GW, Hu YH, Wang JX, Yang WY, An ZX, Hu ZX, Lin J, Xiao JZ, Cao HB, Liu PA, Jiang XG, Jiang YY, Wang JP, Zheng H, Zhang H, Bennett PH, Howard BV. Effects of diet and exercise in preventing NIDDM in people with impaired glucose tolerance. The Da Qing IGT and Diabetes Study. Diabetes Care. 1997 Apr;20(4):537-44. doi: 10.2337/diacare.20.4.537. PMID 9096977
- [Background] American Diabetes Association. Standards of medical care in diabetes--2012. Diabetes Care. 2012 Jan;35 Suppl 1(Suppl 1):S11-63. doi: 10.2337/dc12-s011. No abstract available. PMID 22187469